CLINICAL TRIAL: NCT05369299
Title: Clinical Outcome of Two-piece Zirconia Implants in Immediate Implant Placement - a Prospective Randomized Controlled Clinical Trial
Brief Title: Clinical Outcome of Two-piece Zirconia Implants in Immediate Implant Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIP Ti Zr
Record Dates: First submitted 2022-03-30; First posted 2022-05-11 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Immediate Implantation of Two-piece Zirconia Dental Implants
Keywords: zirconium oxide; Dental Implants; Prospective Studies; Osseointegration; Resonance Frequency Analysis; Patient Reported Outcome Measures; Esthetics

STUDY DESIGN:
Intervention Model Description: prospective controlled randomized trial
Who Masked: Outcomes Assessor
Masking Description: Masking procedures are only applicable for the outcomes assessor. Due to the different colors of the compared implants, blinding procedures are not applicable for the investigator or the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two-piece zirconia implants (Experimental): Immediate dental implant placement will be performed by using the new two-piece zirconia implant Straumann® Pure Ceramic Two Piece Implant
  Interventions: Device: Implant Straumann® Pure Ceramic Two Piece Implant
- Two-piece titanium implants (Active Comparator): Immediate dental implant placement will be performed by using the conventional two-piece titanium implant Neoss® ProActive Tapered Implant
  Interventions: Device: two-piece titanium implant Neoss® ProActive Tapered Implant

INTERVENTIONS:
Device: Implant Straumann® Pure Ceramic Two Piece Implant — Dental implants are placed directly after tooth extraction in the extraction socket.
  Arms: Two-piece zirconia implants
Device: two-piece titanium implant Neoss® ProActive Tapered Implant — Dental implants are placed directly after tooth extraction in the extraction socket.
  Arms: Two-piece titanium implants

SUMMARY:
The purpose of the study is to test whether a two-piece zirconia implant is as reliable in the indication of immediate implant placement as a standard titanium implant.

ELIGIBILITY:
Inclusion Criteria:

Patients giving informed consent to participate in the clinical trial and fulfil the following criteria will be included in the investigation:

1. good oral hygiene standard;
2. good general health;
3. 18 years or older;
4. non-smokers;
5. presence of single-tooth or multiple gaps in the mandible or the maxilla;
6. intact facial bone wall;
7. sufficient bone volume to support an implant of at least 10 mm length.
8. Teeth with removable periapical lesions are included.

Exclusion Criteria:

Primary exclusion criteria are as follows:

1. parafunctional habits;
2. active periodontitis;
3. smoking;
4. pregnancy;
5. acute or chronic medical conditions for which implant therapy has always been considered a contraindication: uncontrolled diabetes (HbA1c >8.0%), mucosal disease, untreated periodontitis, immunological disorders, active malignancy, alcoholism, condition after radiation therapy to the head and neck area and antiresorptive therapy.

   Secondary exclusion criteria will be applied at surgical procedure:
6. loss of facial bone wall due to extraction procedure;
7. insufficient primary stability (less than 32Ncm insertion torque).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Change of PTV | initial, 6 and 12 months after surgical procedure
  Periotest value, Damping capacity assessment. For Periotest values, a customizable healing abutment will be inserted to assess damping capacity.
Change of ISQ | initial, 6 and 12 months after surgical procedure
  Implant stability quotient. A transducer (smart-peg sensor) will be installed on the top of the implant to measure ISQ with resonance frequency analysis. ISQ will be measured from 4 different sites (facial, lingual, mesial, distal) and calculated as mean of measurements.

SECONDARY OUTCOMES:
Change of marginal bone loss | 6 and 12 months after surgical procedure
  A single radiography in paralleling technique will be performed to measure marginal bone loss in millimeters (mm). Individualized x-ray holders will be used to ensure standardization and comparability in radiographic procedure.
Change of PES | 6 and 12 months after surgical procedure
  In the anterior region (4-4) the pink esthetic score (PES) (Fürhauser et al. 2005) will be used to evaluate the esthetic outcome of the soft tissue around the implant-supported single crowns by awarding seven points for the mesial and distal papilla, soft- tissue level, contour, colour, texture and alveolar process deficiency.
Change of width of keratinized mucosa | initial, 12 months after surgical procedure
  The width of keratinized mucosa will be measured in millimetres at the narrowest distance between the mucosal margin and the mucogingival junction at the buccal aspect of the implant using Lugol ́s iodine solution.
Change of BOP | initial, 6 and 12 months after surgical procedure
  Bleeding on probing will be recorded as positive (BOP+) when bleeding of the peri-implant mucosa is detected at implant (tooth) site-level after probing depth assessment within periodontal status.
Gingival biotype | initial
  The tissue phenotype/gingival biotype will be classified at first visit with a conventional periodontal probe. Phenotype will be classified as thin, if the outline of the underlying probe can be seen shining through the buccal mucosa and as thick phenotype, if not.
Mean insertion time | at time of surgery
  Time of implant insertion in seconds (sec).
Change of PROM | initial, 12 months after surgical procedure
  Patient related outcome measures. Patients ́ oral-health related quality of life will be assessed before and 12 months after implant therapy by using a 14-point standardized questionnaire (OHIP-14).
Complications - biological | at time of surgical procedure, 2 weeks, 6 months and 12 months after surgical procedure
  Appearance of biological complications will be recorded in writing. Biological implant complications present the inflammatory reactions on peri-implant tissues, including peri-implant mucositis, peri-implantitis and implant loss.
Complications - biological | at time of surgical procedure
  Appearance of biological complications will be recorded in writing. Biological implant complications present the inflammatory reactions on peri-implant tissues, including peri-implant mucositis, peri-implantitis and implant loss.
Complications - biological | 2 weeks
  Appearance of biological complications will be recorded in writing. Biological implant complications present the inflammatory reactions on peri-implant tissues, including peri-implant mucositis, peri-implantitis and implant loss.
Complications - biological | 6 months
  Appearance of biological complications will be recorded in writing. Biological implant complications present the inflammatory reactions on peri-implant tissues, including peri-implant mucositis, peri-implantitis and implant loss.
Complications - biological | 12 months
  Appearance of biological complications will be recorded in writing. Biological implant complications present the inflammatory reactions on peri-implant tissues, including peri-implant mucositis, peri-implantitis and implant loss.
Complications - technical | at time of surgical procedure
  Appearance of technical complications will be recorded in writing. Technical complications as abutment screw fractures, fractures or chipping of prosthetics may appear due to biomechanical overloading and will be recorded.
Complications - technical | 2 weeks
  Appearance of technical complications will be recorded in writing. Technical complications as abutment screw fractures, fractures or chipping of prosthetics may appear due to biomechanical overloading and will be recorded.
Complications - technical | 6 months
  Appearance of technical complications will be recorded in writing. Technical complications as abutment screw fractures, fractures or chipping of prosthetics may appear due to biomechanical overloading and will be recorded.
Complications - technical | 12 months after surgical procedure
  Appearance of technical complications will be recorded in writing. Technical complications as abutment screw fractures, fractures or chipping of prosthetics may appear due to biomechanical overloading and will be recorded.
Complications - esthetic | at time of surgical procedure
  Appearance of esthetic complications will be recorded in writing. Gingival recession or lack of interdental papillae account for implant esthetic complications and will be recorded.
Complications - esthetic | 2 weeks
  Appearance of esthetic complications will be recorded in writing. Gingival recession or lack of interdental papillae account for implant esthetic complications and will be recorded.
Complications - esthetic | 6 months
  Appearance of esthetic complications will be recorded in writing. Gingival recession or lack of interdental papillae account for implant esthetic complications and will be recorded.
Complications - esthetic | 12 months after surgical procedure
  Appearance of esthetic complications will be recorded in writing. Gingival recession or lack of interdental papillae account for implant esthetic complications and will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Polansky, DMD, Principal Investigator — Department of Dentistry and Oral Health, Medical University of Graz
Locations (1):
- Private practice Prof. Polansky, Graz, Styria, Austria